CLINICAL TRIAL: NCT04485949
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase 2b Study to Assess the Safety and Efficacy of IGV-001, an Autologous Cell Immunotherapy With Antisense Oligonucleotide (IMV-001) Targeting IGF-1R, in Newly Diagnosed Patients With Glioblastoma
Brief Title: A Phase 2b Clinical Study With a Combination Immunotherapy in Newly Diagnosed Patients With Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imvax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14379-201
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: Newly Diagnosed
MeSH Terms: conditions — Glioblastoma | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IGV-001 (Experimental): Participants will be implanted with biodiffusion chambers containing IGV-001 on Day 1 and explanted on Day 3 (at approximately 48 hours following implantation). After 6 weeks, participants will receive radiotherapy (RT) per institutional standards for 5 days per week along with temozolomide 75 mg/m^2 orally, once daily (QD) for up to 12 weeks followed by temozolomide 150 to 200 mg/m^2, orally, on Days 1 to 5 of each 28-day cycle for up to 6 cycles (Week 41).
  Interventions: Combination Product: IGV-001 Cell Immunotherapy; Procedure: Standard of Care (SOC): Radiation Therapy; Drug: SOC: Temozolomide
- Placebo (Placebo Comparator): Participants will be implanted with biodiffusion chambers containing placebo on Day 1 and explanted on Day 3 (at approximately 48 hours following implantation). After 6 weeks, participants will receive RT per institutional standards for 5 days per week along with temozolomide 75 mg/m^2 orally, QD for up to 12 weeks followed by temozolomide 150 to 200 mg/m^2, orally, on Days 1 to 5 of each 28-day cycle for up to 6 cycles (Week 41).
  Interventions: Combination Product: Placebo; Procedure: Standard of Care (SOC): Radiation Therapy; Drug: SOC: Temozolomide

INTERVENTIONS:
Combination Product: IGV-001 Cell Immunotherapy — IGV-001, an immunotherapeutic product that combines personalized whole tumor-derived cells with an antisense oligonucleotide (IMV-001) in implantable biodiffusion chambers.
  Arms: IGV-001
Combination Product: Placebo — Placebo in implantable biodiffusion chambers containing a predetermined inactive solution.
  Arms: Placebo
Procedure: Standard of Care (SOC): Radiation Therapy — Radiation therapy administered per institutional standards.
Drug: SOC: Temozolomide — Temozolomide administered orally.

SUMMARY:
The purpose of this study is to assess progression-free survival (PFS) and overall survival (OS) in newly diagnosed Glioblastoma (GBM) participants treated with IGV-001 as compared with placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a Karnofsky performance scale (KPS) score ≥ 70 at screening
* Has a new diagnosis of GBM (WHO GRADE III or Grade IV GBM) based on the treating neurosurgeon's best clinical judgement
* Has a diagnostic contrast-enhanced magnetic resonance imaging (MRI) scan with fluid attenuated inversion-recovery (FLAIR) sequence of the brain at screening. Participants must have a confirmed measurable disease pre-operatively with at least 1 lesion measuring a total bi-perpendicular product of 4 centimeter square (cm^2) in 2 different planes (axial, sagittal, or coronal)
* The tumor must be located in the supratentorial compartment
* Has adequate bone marrow and organ function at screening

Key Exclusion Criteria:

* Has bi-hemispheric disease, multicentric disease, or disease burden involving the brain stem or cerebellum based on MRI post-gadolinium enhancement
* Has received any previous surgical resection or any anticancer intervention for glioma
* Has any history of glioma, a concurrent malignancy, or malignancy within 3 years of randomization, unless definitive therapy is completed, with the exception of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has completed curative therapy
* Has any severe immunocompromised condition (eg, human immunodeficiency virus (HIV) with a cluster of differentiation [CD] 4+ cell count <200*10^6/liter [L]) or any active uncontrolled autoimmune disease (eg, Crohn's disease)
* Has an active cardiac disease or a history of cardiac dysfunction
* Is receiving any other investigational agent(s) or has received an investigational agent within 30 days or 5 half-lives of investigational agent use, whichever is longer, prior to screening
* Is partaking in another interventional study. Participants who are partaking in an observational study are eligible
* Has received a live vaccine within 30 days of screening
* Has active and uncontrolled/untreated hepatitis B virus (HBV), hepatitis C virus (HCV), HIV, or any other active infections that, in the Investigator's opinion, would impair or prohibit a participant's participation in this study.
* Is receiving treatment with Tumor Treating Fields or Optune®

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 36 months
  PFS is defined as the time from randomization to first progression, as determined by the central radiology review group blinded to the study treatment arm, or death.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 48 months
  OS is defined as the time from randomization to death due to any cause.
Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Events (ADE), and Unexpected Adverse Device Events (ADR) | Up to 36 months
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a product, which does not have a causal relationship with treatment. AEs will be graded according to Common Terminology Criteria for Adverse Events, version 5.0 from mild(Grade 1) to death(Grade 5). SAE is an AE which is considered serious if it results in any of the following outcomes: death, life-threatening AE, require hospitalizations/prolongation of hospitalizations, results in persistent or significant disability; results in a congenital anomaly and is a medically important event. An ADE is defined as any AE caused by or associated with use of a device and suspected to be resulting from insufficiencies in the instructions for use, the deployment, the implantation, the installation, the operation, or any malfunction of the medical device. An Unexpected ADR is defined as an adverse reaction, nature or severity of which is not consistent with product information.
Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to 36 months
Number of Participants With Clinically Significant Vital Signs Measurements | Up to 36 months
Number of Participants With Clinically Significant Physical Examination Findings | Up to 36 months

OTHER OUTCOMES:
Time to Deterioration of Karnofsky Performance Status (KPS) Score | Up to 36 months
  Time to KPS deterioration is defined as the time from screening to the first date of deterioration of the KPS score. Deterioration of KPS is defined as a stable or increasing steroid dose-dependent stabilization of a KPS score of <70 over 2 consecutive visits at least 4 weeks apart. KPS is an 11-level score which ranges between 0 (death) to 100 (complete healthy status); a higher score represents a higher ability to perform daily tasks.
PFS in Participants With O6-methylguanine-DNA Methyltransferase (MGMT) With Methylation [MGMT+] and MGMT Without Methylation [MGMT-] | Up to 36 months
  PFS is defined as the time from randomization to first progression, as determined by the central radiology review group blinded to the study treatment arm, or death. MGMT status will be determined per epigenetic and tumor proliferation analysis from tissue obtained during surgery.
OS in Participants With MGMT+ and MGMT- | Up to 48 months
  OS is defined as the time from randomization to death due to any cause. MGMT status will be determined per epigenetic and tumor proliferation analysis from tissue obtained during surgery.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northwell Health at North Shore University Hospital, Manhasset, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - UC Health, Cincinnati, Ohio
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee IY, Hanft S, Schulder M, Judy KD, Wong ET, Elder JB, Evans LT, Zuccarello M, Wu J, Aulakh S, Agarwal V, Ramakrishna R, Gill BJ, Quinones-Hinojosa A, Brennan C, Zacharia BE, Silva Correia CE, Diwanji M, Pennock GK, Scott C, Perez-Olle R, Andrews DW, Boockvar JA. Autologous cell immunotherapy (IGV-001) with IGF-1R antisense oligonucleotide in newly diagnosed glioblastoma patients. Future Oncol. 2024 Mar;20(10):579-591. doi: 10.2217/fon-2023-0702. Epub 2023 Dec 7. PMID 38060340
- [Derived] Andrews CE, Zilberberg J, Perez-Olle R, Exley MA, Andrews DW. Targeted immunotherapy for glioblastoma involving whole tumor-derived autologous cells in the upfront setting after craniotomy. J Neurooncol. 2023 Dec;165(3):389-398. doi: 10.1007/s11060-023-04491-4. Epub 2023 Nov 29. PMID 38017340